CLINICAL TRIAL: NCT02578914
Title: A Randomized, Parallel, Single-Center, Double-Masked, Vehicle-Controlled Phase II Study to Evaluate the Activity of NS2 Ophthalmic Solution in Subjects With Allergic Conjunctivitis Using the Conjunctival Allergen Provocation Test (CAPT)
Brief Title: A Safety and Activity Study of NS2 in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALDNS2-203-D1; 15-MO-001 (Other: Aldeyra Therapeutics Inc.)
Record Dates: First submitted 2015-10-08; First posted 2015-10-19 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2016-05

CONDITIONS: Allergic Conjunctivitis; Seasonal Allergies
Keywords: allergic conjunctivitis; seasonal allergies; ragweed allergy; grass allergy; tree allergy; NS2; Aldeyra
MeSH Terms: conditions — Conjunctivitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NS2 Ophthalmic Drops (0.5%) (Experimental): NS2 Ophthalmic Drops (0.5%)
  Interventions: Drug: NS2 Ophthalmic Drops (0.5%)
- NS2 Ophthalmic Drops Vehicle (0.0%) (Sham Comparator): NS2 Ophthalmic Drops Vehicle (0.0%) control
  Interventions: Drug: NS2 Ophthalmic Drops Vehicle (0.0%)

INTERVENTIONS:
Drug: NS2 Ophthalmic Drops (0.5%)
  Arms: NS2 Ophthalmic Drops (0.5%)
Drug: NS2 Ophthalmic Drops Vehicle (0.0%)
  Arms: NS2 Ophthalmic Drops Vehicle (0.0%)

SUMMARY:
This is a randomized, parallel, single center, double masked, vehicle controlled study. The purpose of this study is to determine the activity and safety of NS2 in patients with grass, tree or ragweed-pollen induced seasonal allergic conjunctivitis . Subjects will be randomized 1:1 to receive multiple doses of NS2 Ophthalmic Drops (0.5%) or NS2 Ophthalmic Drops Vehicle (0.0%).

Free aldehydes are thought to be related to inflammatory conditions such as allergic conjunctivitis. NS2, a small molecule aldehyde trap, is being evaluated to determine whether it may decrease inflammation by lowering aldehyde levels.

ELIGIBILITY:
Inclusion Criteria:

* Graded conjunctival redness in at least one region (nasal or temporal) in each eye at any one time point (not necessarily the same time point) post-CAPT (Conjunctival Allergen Provocation Test) of >2
* Graded ocular itching at any one time point
* Visual acuity of at least 20/50 in each eye
* At least 2 year history of moderate to severe allergic conjunctivitis.
* Positive skin prick test to ragweed, grass and/or tree pollen within one year of Screening Visit (Visit 1).
* Ability to avoid any topical or systemic ocular medications during the entire study period.

Exclusion Criteria:

* Subjects must not have an ocular itching score >0 or a conjunctival redness score >1 prior to CAPT in either eye in any region (nasal or temporal) at Visits 2-4. I
* History of glaucoma, or Intraocular Pressure (IOP) over 25mmHg at the screening visit, or a history of elevated IOP within the past 1 year.
* Ocular surgery, including laser procedures, within the past 12 months of Visit 1.
* Use of glaucoma medications, antibiotics, antivirals, or topical cyclosporine within 1 month of the screening visit.
* History of dry eye syndrome, blepharitis, herpes simplex keratitis or herpes zoster keratitis.
* History of uveitis in the past 3 years.
* Presence of any ocular infection or active ocular inflammation (e.g. follicular conjunctivitis, allergic conjunctivitis) within 14 days prior to start of study (Visit 1).
* History of moderate to severe asthma or allergy induced asthma to the allergen that will be used in CAPT.
* Use of oral corticosteroids within 30 days of screening and throughout the study period; use of intranasal or inhaled corticosteroids within 14 days of screening and throughout the study period.
* Use of antihistamines (ocular, nasal, topical or oral) within 7 days prior to screening (Visit 1) and throughout the study period. Non-medicated artificial tears are allowed up to 72 hours before screening (Visit 1) and throughout the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, Principal Investigator — Inflamax Research Incorporated
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- NS2 Ophthalmic Drops (0.5%): NS2 administered QID (four times daily) for approximately 2 weeks
- Vehicle Ophthalmic Drops: Vehicle administered QID for approximately 2 weeks
Period: Overall Study
Arm/Group | NS2 Ophthalmic Drops (0.5%) | Vehicle Ophthalmic Drops
Started | 50 | 50
Completed | 48 | 50
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- NS2 Ophthalmic Drops (0.5%): NS2 administered QID for approximately 2 weeks
- Total: Total of all reporting groups
Arm/Group | NS2 Ophthalmic Drops (0.5%) | Vehicle Ophthalmic Drops | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.5) | 41.9 (12.1) | 43.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 56
  Male | 18 | 26 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 45 | 45 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 9 | 22
  Black or African American | 11 | 8 | 19
  Native Hawaiian / other Pacific Islander | 0 | 0 | 0
  White | 22 | 30 | 52
  Other | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Score at Day 14, 60 Minutes Into the Allergen Challenge
Description: Mean change from baseline in ocular itching score using a 0 to 4 scale (0 = none, 4 = severe) on Day 14, 60 minutes into the allergen challenge. The least squares mean (standard error) was derived from analysis of covariance (ANCOVA) with baseline as a covariate and treatment group as a factor.
Time Frame: The efficacy assessment period was assessed at Day 14; baseline was Day -7.
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NS2 Ophthalmic Drops (0.5%) | Vehicle Ophthalmic Drops
Number analyzed (Participants) | 50 | 50
units on a scale | -1.550 (0.168) | -1.013 (0.163)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject was approximately 9 weeks.
Arm/Group | NS2 Ophthalmic Drops (0.5%) | Vehicle Ophthalmic Drops
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 49/50 | 11/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NS2 Ophthalmic Drops (0.5%) (N=50) | Vehicle Ophthalmic Drops (N=50)
General disorders and administration site conditions (General disorders) | 49 | 4 — Transient and self-limiting instillation site irritation that resolved in all cases.
Lacrimination increased (Eye disorders) | 3 | 0
Punctate keratitis (Eye disorders) | 3 | 2
Headache (Nervous system disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes